CLINICAL TRIAL: NCT02355964
Title: EFFORT Asthma: Effects of a High Protein/Low Glycemic Index Diet and Physical Exercise in Sedentary Non-obese Asthmatics.
Brief Title: EFFORT Asthma: Effects of Diet and Exercise in Asthma
Acronym: EFFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Louise Lindhardt Toennesen, MD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFFORT Asthma
Record Dates: First submitted 2015-01-16; First posted 2015-02-04 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- exercise (Experimental): exercise (Aerobe training) 3 times per week
  Interventions: Behavioral: Exercise
- Diet (Experimental): A diet with an overall high protein content and a low glycemic index
  Interventions: Behavioral: Diet
- Diet+Exercise (Experimental): A diet with an overall high protein content and a low glycemic index combined with exercise (Aerobe training) 3 times per week.
  Interventions: Behavioral: Exercise; Behavioral: Diet
- control (No Intervention): Regular lifestyle (no intervention)

INTERVENTIONS:
Behavioral: Exercise — Aerobe exercise 3 times a week in 8 weeks
  Arms: Diet+Exercise; exercise
Behavioral: Diet — Diet (a diet with an overall high protein content and a low glycemic index) in 8 weeks
  Arms: Diet; Diet+Exercise

SUMMARY:
This project aims to study the effects of lifestyle changes on asthma and systemic inflammation in a randomized clinical trial of diet and exercise. The project is a multidisciplinary collaboration in the areas of medicine, physiology and nutrition, centred on improving asthma control in non-obese sedentary asthmatics via simple means.

DETAILED DESCRIPTION:
After screening and enrollment, a total of 200 Danish sedentary, non-obese asthma patients will be randomized to one of four groups: 1) control group (no intervention), 2) physical exercise intervention, 3) diet intervention (a diet with an overall high content of protein and a low glycemic index) or 4) exercise plus diet intervention.

Asthma is defined as respiratory symptoms and at least one positive asthma test. Patients will continue their regular doses of anti-asthma treatment unchanged throughout the study period. Type of anti-inflammatory medicine will be recorded and the adherence to the therapy will be assessed before the intervention period and at follow-up using questionnaires

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Uncontrolled or partly uncontrolled asthma
* Capable of exercising on bike
* Sedentary (currently do less than 60 min of structured/planned physical activity per week)

Exclusion Criteria:

BMI ≥ 30.0 or <20.5

* Chronic obstructive pulmonary disease (COPD), pregnancy, other inflammatory or metabolic diseases
* The use of oral anti-inflammatory medication or the use of antibiotic treatment during the last 8 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (Juniper) (ACQ). | Within 10 days (+/- 1 day) of completing the intervention

SECONDARY OUTCOMES:
Airway hyperresponsiveness to mannitol, as measured by an airway provocation test. | Within 10 days (+/- 1 day) of completing the intervention
  The response-dose-ratio (RDR) will be calculated as the percentage fall in forced expiratory volume in 1 second (FEV1) after the last dose of inhaled dried mannitol powder delivered, divided by the cumulative dose of inhaled mannitol.
Systemic low-grade inflammation, as measured by serum-levels (in microgram/ml) of high sensitivity C-reactive protein, interleukin 6 (IL-6), IL-8, tumor necrosis factor alpha (TNF-alpha) and leptin. | Within 10 days (+/- 1 day) of completing the intervention
Fractional exhaled nitric oxide (FeNO) | Within 10 days (+/- 1 day) of completing the intervention
  FeNO (a marker of eosinophilic inflammation)
Sputum inflammatory cell count | Within 10 days (+/- 1 day) of completing the intervention
  Number and type of inflammatory cells in induced sputum
Adipose tissue inflammatory properties as measured by levels of messenger ribonucleic acid (mRNA) of IL-6, IL-8, leptin and TNF-alpha in abdominal fat biopsies. | Within 10 days (+/- 1 day) of completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Professor, Study Chair — Respiratory Research Unit, Bispebjerg hospital
Locations (1):
- Respiratory Research Unit, Birpebjerg Hospital, Copenhagen NV, Denmark